CLINICAL TRIAL: NCT00057746
Title: A Phase II Randomized Trial Of Two Dose Schedules For Delivering Prophylactic Cranial Irradiation For Patients With Limited Disease Small Cell Lung Cancer
Brief Title: Brain Irradiation in Treating Patients With Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0212; CDR0000258668
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Active Comparator): Prophylactic cranial irradiation, 2.5 Gy fx
  Interventions: Radiation: Prophylactic cranial irradiation, 2.5 Gy fx
- Arm II (Experimental): Prophylactic cranial irradiation, 2.0 Gy fx
  Interventions: Radiation: Prophylactic cranial irradiation, 2.0 Gy fx
- Arm III (Experimental): Prophylactic cranial irradiation, 1.5 Gy fx
  Interventions: Radiation: Prophylactic cranial irradiation, 1.5 Gy fx

INTERVENTIONS:
Radiation: Prophylactic cranial irradiation, 2.5 Gy fx — Prophylactic cranial irradiation, 2.5 Gy once daily, M-F, in 10 fractions (fx) for a total of 25 Gy
  Other Names: PCI
  Arms: Arm I
Radiation: Prophylactic cranial irradiation, 2.0 Gy fx — Prophylactic cranial irradiation, 2.0 Gy once daily, M-F, in 18 fractions (fx) for a total of 36 Gy
  Other Names: PCI
  Arms: Arm II
Radiation: Prophylactic cranial irradiation, 1.5 Gy fx — Prophylactic cranial irradiation, 1.5 Gy twice daily, M-F, in 24 fractions (fx) for a total dose of 36 Gy
  Other Names: PCI
  Arms: Arm III

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known which radiation therapy regimen is more effective in preventing brain metastases in patients with limited-stage small cell lung cancer while taking into account chronic neurotoxicity from radiation therapy.

PURPOSE: This randomized phase II trial compares the incidence of chronic neurotoxicity between three different brain irradiation regimens. The corresponding phase III component addressing the prevention of brain metastases was run by EORTC and reported separately (NCT00005062).

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the incidence of chronic neurotoxicity in patients treated with these regimens.
* Compare quality of life of patients treated with these regimens. (phase III closed to accrual as of 12/31/05)

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (60 and under vs over 60) and time since induction therapy (90 days or less vs 91-180 days vs 181-240 days). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients undergo prophylactic cranial irradiation (PCI) once daily 5 days a week. Treatment continues for 2 weeks in the absence of unacceptable toxicity.
* Arm II: Patients undergo PCI once daily 5 days a week. Treatment continues for 2.6 weeks in the absence of unacceptable toxicity.
* Arm III: Patients undergo PCI twice daily 5 days a week. Treatment continues for 3.4 weeks in the absence of unacceptable toxicity.

Quality of life is assessed at baseline, every 6 months for 1 year, and then annually for 3 years.

Patients are followed every 6 months for 1 year and then annually for 3 years.

PROJECTED ACCRUAL: A total of 264 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer by fine needle aspiration, biopsy, or 2 positive sputa

  * Limited stage (I-IIIB)

    * Confined to 1 hemithorax
    * No T4 based on malignant pleural effusion, or N3 disease based on contralateral hilar or contralateral supraclavicular involvement
* Complete response after induction chemotherapy (with or without thoracic radiotherapy)
* Consolidative chest radiotherapy may be initiated before study
* No radiographic evidence of any of the following:

  * Brain metastases

    * Normal brain CT scan or MRI less than 1 month before study
  * Ipsilateral lung metastases
  * Malignant pleural effusion

    * Minimal pleural effusion by chest CT scan allowed, but not by chest x-ray

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin at least 10.0 g/dL^

Hepatic

* Not specified

Renal

* Not specified

Pulmonary

* See Disease Characteristics

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Neurological function class 1 or 2
* No epilepsy requiring permanent oral medication
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other serious medical or psychiatric condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* At least 1 week since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior external beam radiotherapy to the head or neck, including stereotactic radiotherapy
* Concurrent thoracic radiotherapy allowed

Surgery

* Not specified

Other

* No concurrent antitumor agents

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2003-02; Primary Completion 2009-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron H. Wolfson, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (222):
- United States (217):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Osborn, Scottsdale, Arizona
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Shea, Scottsdale, Arizona
  - Highlands Oncology Group - Springdale, Springdale, Arkansas
  - Auburn Radiation Oncology, Auburn, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Bay Medical, Panama City, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis, Indianapolis, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - South Suburban Oncology Center, Quincy, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Immanuel St. Joseph's, Mankato, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Cancer Institute of Cape Girardeau, LLC, Cape Girardeau, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Radiation Oncology Associates - Reno, Reno, Nevada
  - Ocean Medical Center at Meridian Health, Brick, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Hudson Valley Oncology Associates, Poughkeepsie, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Huron Hospital Cancer Care Center, Cleveland, Ohio
  - Euclid Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - South Pointe Hospital Cancer Care Center, Warrensville Heights, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Cancer Center at PMCC, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center CCOP Research Base, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Arlington Cancer Center - Arlington, Arlington, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - St. Joseph Cancer Center, Bellingham, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
- Canada (5):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - McGill Cancer Centre at McGill University, Montreal

REFERENCES:
- [Background] Gondi V, Paulus R, Bruner D, et al.: Prognostic significance of QOL deterioration during early lung cancer survivorship: secondary analysis of RTOG 0212 and 0214. [Abstract] J Clin Oncol 29 (Suppl 15): A-6061, 2011.
- [Background] Le Pechoux C, Dunant A, Senan S, Wolfson A, Quoix E, Faivre-Finn C, Ciuleanu T, Arriagada R, Jones R, Wanders R, Lerouge D, Laplanche A; Prophylactic Cranial Irradiation (PCI) Collaborative Group. Standard-dose versus higher-dose prophylactic cranial irradiation (PCI) in patients with limited-stage small-cell lung cancer in complete remission after chemotherapy and thoracic radiotherapy (PCI 99-01, EORTC 22003-08004, RTOG 0212, and IFCT 99-01): a randomised clinical trial. Lancet Oncol. 2009 May;10(5):467-74. doi: 10.1016/S1470-2045(09)70101-9. Epub 2009 Apr 20. PMID 19386548
- [Background] Pechoux CL, Hatton M, Kobierska A, et al.: Randomized trial of standard dose to a higher dose prophylactic cranial irradiation (PCI) in limited-stage small cell cancer (SCLC) complete responders (CR): primary endpoint analysis (PCI99-01, IFCT 99-01, EORTC 22003-08004, RTOG 0212). [Abstract] J Clin Oncol 26 (Suppl 15): A-LBA7514, 2008.
- [Result] Wolfson AH, Bae K, Komaki R, Meyers C, Movsas B, Le Pechoux C, Werner-Wasik M, Videtic GM, Garces YI, Choy H. Primary analysis of a phase II randomized trial Radiation Therapy Oncology Group (RTOG) 0212: impact of different total doses and schedules of prophylactic cranial irradiation on chronic neurotoxicity and quality of life for patients with limited-disease small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2011 Sep 1;81(1):77-84. doi: 10.1016/j.ijrobp.2010.05.013. Epub 2010 Aug 26. PMID 20800380

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Prophylactic cranial irradiation, 2.5 Gy FX: Prophylactic cranial irradiation, 2.5 Gy once daily, M-F, in 10 fractions for a total of 25 Gy
- Arm II: Prophylactic cranial irradiation, 2.0 Gy FX: Prophylactic cranial irradiation, 2.0 Gy once daily, M-F, in 18 fractions for a total of 36 Gy
- Arm III: Prophylactic cranial irradiation, 1.5 Gy FX: Prophylactic cranial irradiation, 1.5 Gy twice daily, M-F, in 24 fractions for a total dose of 36 Gy
Period: Overall Study
Arm/Group | Arm I | Arm II | Arm III
Started | 131 | 67 | 67
Completed | 131 | 67 | 66
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Arm III | Total
Number analyzed (Participants) | 131 | 67 | 66 | 264
Age, Continuous [Median (Full Range); unit: years] | 62 [39 to 86] | 62 [39 to 78] | 61 [44 to 77] | 62 [39 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 33 | 32 | 118
  Male | 78 | 34 | 34 | 146

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Chronic Neurotoxicity
Description: Chronic neurotoxicity is defined as a drop in one standard error of measurement (SEM) in any one of the three tests comprising the neuropsychological test battery (Hopkins Verbal Learning Test, Controlled Word Association Test, and Trail-Making Test) without development of brain metastasis by one year. The SEM is calculated as the standard deviation of the baseline test multiplied by the square root of one minus the published reliability coefficient for the test.
Time Frame: From study registration to one year.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 45 | 20 | 19
percentage of participants | 60 [48 to 72] | 85 [72 to 98] | 89 [78 to 100]

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-serious adverse events.
Arm/Group | Arm I | Arm II | Arm III
Serious Adverse Events (participants affected / at risk) | 6/128 | 2/66 | 4/64
Other Adverse Events (participants affected / at risk) | 54/128 | 37/66 | 26/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=128) | Arm II (N=66) | Arm III (N=64)
Abdominal pain or cramping (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia-esophageal related to radiation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Constitutional Symptoms - Other, Specify (General disorders) | 0 | 0 | 1
Edema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0
Weight loss (Investigations) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic/laboratory-Other (Metabolism and nutrition disorders) | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain (Nervous system disorders) | 0 | 0 | 1
Confusion (Nervous system disorders) | 1 | 0 | 0
Neuropathy - motor (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Vertigo (Nervous system disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=128) | Arm II (N=66) | Arm III (N=64)
Nausea or vomiting (Gastrointestinal disorders) | 21 | 18 | 11
Fatigue (General disorders) | 35 | 25 | 17
Headache (Nervous system disorders) | 31 | 21 | 19
Insomnia (Psychiatric disorders) | 5 | 4 | 4

LIMITATIONS AND CAVEATS:
The number of inevaluable patients at one year (e.g., patients dying prior to 1 year, patients not completing the neurocognitive battery at 1 year) was greater than anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.